CLINICAL TRIAL: NCT03534765
Title: Frailty and Sarcopenia Outcomes in Emergency General Surgery
Acronym: FrOGS
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Yeovil District Hospital NHS Foundation Trust (Other)
Collaborators: University Hospital Southampton NHS Foundation Trust (Other); Basingstoke and North Hampshire Hospital (Unknown); Dorset County Hospital NHS Foundation Trust (Other Government); Poole Hospital NHS Foundation Trust (Other); Portsmouth Hospitals NHS Trust (Other Government); Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust (Other Government); Salisbury NHS Foundation Trust (Other Government); University of Southampton (Other); National Institute for Health Research, United Kingdom (Other Government); Hampshire Hospitals NHS Foundation Trust (Other); Isle of Wight NHS Trust (Other)
Responsible Party: Principal Investigator, Nathan Curtis, Clinical Research Fellow, Yeovil District Hospital NHS Foundation Trust
Other Study IDs: 224891
Record Dates: First submitted 2018-03-27; First posted 2018-05-23 (Actual); Last update posted 2019-01-10 (Actual); Status verified 2019-01

CONDITIONS: Frail Elderly Syndrome; Emergencies; Surgery; Sarcopenia
Keywords: Laparotomy; Frailty; Sacropenia
MeSH Terms: conditions — Emergencies; Sarcopenia; Frailty

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Retrospective arm: Retrospective multicentre cohort with 1 year outcomes available following emergency surgery for NELA eligible gastrointestinal pathology. Please refer to WP1 inclusion and exclusion criteria for eligibility.
  Interventions: Diagnostic Test: CT abdomen +/- pelvis; Procedure: Emergency laparotomy for general surgical pathology
- Prospective, multicentre arm: 10 centre prospective observational arm. Please refer to WP2 inclusion and exclusion criteria for eligibility.
  Interventions: Diagnostic Test: CT abdomen +/- pelvis; Diagnostic Test: Edmunton Frailty Score; Procedure: Emergency laparotomy for general surgical pathology

INTERVENTIONS:
Diagnostic Test: CT abdomen +/- pelvis — Diagnostic CT scan (only if requested by responsible clinicians)
Diagnostic Test: Edmunton Frailty Score — Patient completed previously valided questionnaire quantifying frailty.
  Groups: Prospective, multicentre arm
Procedure: Emergency laparotomy for general surgical pathology — Emergency general surgical laparotomy (defined by the UK NELA body)

SUMMARY:
1. A retrospective scoping cohort review of adult patients undergoing emergency laparotomy/laparoscopy for acute gastrointestinal (GI) pathology who have had a CT scan of the abdomen(+/- pelvis). CT measured sarcopenia would be compared with clinical outcomes, 30-day and 1-year mortality.
2. A prospective observational cohort study and bio-banking exercise of routinely collected clinical data, in a cohort of patient undergoing emergency laparotomy/laparoscopy or conservative treatment for an otherwise operable pathology. An interrogation of CT measured sarcopenia and a validated clinical frailty score would be analysed against clinical outcomes, 30-day and 1-year mortality.

The investigators aim to research the association and predictive advantage of combining subjectively measured frailty, objectively measured CT sarcopenia and other risk predicting tools used in every day surgical practice and surgical outcomes (mortality and morbidity) in a cohort of acute surgical patients undergoing surgery or conservative treatment.

DETAILED DESCRIPTION:
Frailty has a significant impact on surgical outcomes. It is an independent risk factor for adverse outcomes following surgery including complications, length of stay, inability to return home and mortality. Frailty is a physiological decline across multiple body systems accumulating in loss of reserves and increased vulnerability to stressors.

Sarcopenia, loss of muscle mass or progressive reduction in muscle mass, is one of the central physiological manifestations of frailty resulting in weight loss, weakness and exhaustion. Frailty has both a strong correlation with age as well as significant overlap with disability and co-morbidity. Further factors strongly influencing outcome, 30 day and mortality have been described including polypharmacy, Charlson co-morbidity index, age, not independently mobile, emergency admission and falls. It has been recognised that poor outcomes are multimodal relating to the interplay of co-morbidities, physical functioning and nutrition.

Assessing frailty can be completed using simple questionnaire tools, as well as more complex assessment of co-morbidity, functional status, and disability. There is good evidence the simple tools can be as accurate as formal geriatric assessments.

As sarcopenia relates directly to many manifestations of frailty it can be used as a surrogate marker. One of the favoured ways for diagnosing sarcopenia is using CT morphometric biological markers. This uses an axial image at the level of the 3rd lumbar vertebra (L3) to assess the total or cross-sectional volume of the psoas muscle, giving rise to indices measuring muscle mass, visceral adipose tissue and subcutaneous adipose tissue.

Major abdominal emergency surgery is a high-risk procedure with ongoing audit and outcome monitoring. Currently data collection for UK National Emergency Laparotomy Audit (NELA) is in its fourth year with annual reports into the management and outcomes of emergency laparotomies. Observation and audit of these outcomes remain central to improving service and healthcare both regionally and nationally. Furthermore, this group of patients is not well represented in research and is one of the most understudied surgical cohorts that exist. This is especially the case for patients presenting with an acute surgical diagnosis and are deemed unable to withstand the stress of surgery, and hence pursue a conservative or radiological treatment option. With our ageing, co-morbid population this is becoming increasing common. The diagnosis of frailty and sarcopenia are a significant measurable and modifiable risk factor that impacts on perioperative surgical care, healthcare provider and patient decision-making and most importantly long and short term outcomes. This urgently requires further audit and study.

Work package one (WP1): Retrospective scoping cohort study in acute general surgery

Patient identification The number of patients recruited from each participating hospital will be proportionate to the total number of cases, in accordance with relative annual case volumes (as reported by NELA - in the case of less than 100% case capture, the theoretical 100% case number will be used). This will provide a representative sample of the recruiting region's population.

The most recent laparotomy cases with 1-year follow-up mortality data available will be included at the time of study activation. Data collection over a predicted six week period will be undertaken or until the sample size is reached. Retrospective collection of routinely recorded clinical data will be performed (See appendix data collection tool). This includes, but is not restricted to [a] routine clinical variables: patient characteristics, demographic, pathological and physiological variables will be captured in line with NELA data, alongside confounding factors associated with frailty and sarcopenia.

Protocol for measuring muscle radiation attenuation Inclusion: Retrievable CT abdomen/pelvis on an electronic NHS PACS system. CT can be non-contrast or with contrast, supine or prone but must be of sufficient quality for the sarcopenia CT analyses software to handle (Slico-matic™, TomoVision, Magog, Canada ).

Exclusion: CT-scans with large radiation artefacts or with missing parts of muscle tissue on the ventral, dorsal, or both lateral edges of the scan preventing sarcopenia assessment.

Patients meeting inclusion criteria will have their CT extracted and reviewed by a trained independent party. This may through an allocated representative at the base hospital or the CT can be extracted and sent in a fully anonymised format to the central unit for sarcopenia assessment. CT scans obtained via a PACS system can up transferred through secure inter-hospital PACS transfer. Those with non-compatible systems can either be uploaded via CD or analysed at the data collection site. The outcome of the assessment for sarcopenia will define whether a patient is considered to have sarcopenia.

Participants can be identified primarily from the NELA database with confirmation of GI pathology on the radiological report. This can be cross reference against admission logs, acute surgery admission databases, theatre logs for emergency surgery and NELA databases to maximise case capture. Once patients are confirmed to meet the inclusion criteria their data can be gathered into a data collection tool. The CT scan will be extracted and sent for analysis.

All patients meeting inclusion criteria will be identified by the lead researcher in each centre. Frailty scores are already part of standard acute admission clerking proformas in many of the hospitals across the region; as such the researcher's role will be ensure appropriate and complete data capture from existing clinical information sources, but no additional intervention or questioning of patients beyond current standard of care will be required. Patients will be collected across a set time scale as listed above. Baseline demographics and disease factors will be collected as per collection proforma attached as supplementary material.

The Reported Edmonton Frail Scale (REFS) is collected at time of admission as part of routine clinical assessment for surgical admissions. This is a validated, self-reported patient questionnaire that can categorise the degree of frailty. This information is routinely collected in many acute unit or care of the elderly departments. The REFS will enable a consistent method of collecting this data utilising a rapid and well validated tool.

For patients presenting in extremis or unable to complete the score due to an acute state or requirement for prompt treatment, this will be gathered at the next appropriate pre-operative opportunity. Patients unable to complete a REFS given the best opportunity will be excluded, however reasons for exclusion will be recorded.

ELIGIBILITY:
Inclusion Criteria:

* Adults age over 18
* Route of admission should include all general surgical admission or referrals via emergency department, interdepartmental transfers, direct referrals and GP referrals to an acute general surgical team.
* All patients are required to have had a CT scan abdomen or abdomen and pelvis, supine or prone, with or without contrast.
* All patients are required to have a completed REFS.
* Those treated with operative measure (NCEPOD criteria) or those that would be treated operatively as an emergency, expedited, or urgently on the GI tract including:
* Laparoscopic, open, converted or laparoscopic assisted
* Surgical or radiological procedure or conservative treatments for pathology involving the stomach, small bowel, large bowel as a result of perforation, obstruction, ischaemia, bleeding or abscess.
* Washout or evacuation of intrabdominal haematoma or abscess
* Laparotomy or laparoscopy with no intervention due to inoperable pathology where the intention was to perform definition intervention.
* Bowel resection or repair or conservative treatment due to obstructed or incarcerated incisional umbilical femoral or inguinal hernia.
* Bowel resection/repair or conservative treatment due to obstructing/incarcerated incisional hernias provided the presentation and findings were acute. This will include large incisional hernia repair with division of adhesions.
* Laparoscopic/Open Adhesiolysis or conservative treatment for bowel obstruction
* Return to theatre for repair of substantial dehiscence of major abdominal wound (i.e. "burst abdomen")
* Any reoperation/return to theatre or conservative treatment for complications of elective general/upper GI surgery meeting the criteria above is included. Returns to theatre for complications following non-GI surgery are excluded (see exclusion criteria below).
* If multiple procedures are performed on different anatomical sites within the abdominal/pelvic cavity, the patient would be included if the major procedure is general surgical.
* Non-elective colonic resection with hysterectomy for a fistulating colonic cancer would be included as the bowel resection is the major procedure
* Bowel resection at the same time as emergency abdominal aortic aneurysm repair would not be included as the aneurysm repair is the major procedure
* The subjects are required to have had an acute admission, inpatient stay, formal ward admission, review and diagnosis of acute GIT surgical pathology under an acute surgical team.

Exclusion Criteria:

* Do not meet inclusion criteria for specific work package
* Patients less than 18 years old
* Ambulant or day case admission or outpatient admission only
* No review from an acute surgical team.
* Prisoners or patients under arrest or on remand.
* Isolated gynaecology pathology: pathology of the ovaries, uterus or tubal systems not involving the gastrointestinal tract(GIT) i.e ectopic pregnancy.
* Isolated urology acute abdomen: pathology of the kidneys, ureters or bladder not involving the GIT i.e pyelonephritis, lower urinary tract infections, renal or ureteric stones, bladder malignancy
* Isolated vascular pathology I.e Ruptured aortic aneurysm with no GIT ischaemia, iliac aneurysmal disease.
* Excluded uncomplicated appendicectomy, cholecystectomy and ventral wall, or inguinal hernia.
* Elective laparotomy / laparoscopy
* Diagnostic laparotomy/laparoscopy where no subsequent procedure is performed (NB, if no procedure is performed because of inoperable pathology, the case is included).
* Appendicectomy +/- drainage of localised collection unless the procedure is incidental to a non-elective procedure on the GI tract
* Cholecystectomy +/- drainage of localised collection unless the procedure is incidental to a non-elective procedure on the GI tract (All surgery involving the appendix or gallbladder, including any surgery relating to complications such as abscess or bile leak is excluded. The only exception to this is if carried out as an incidental procedure to a more major procedure. We acknowledge that there might be extreme cases of peritoneal contamination, but total exclusion avoids subjective judgement calls about severity of contamination.)
* Non-elective hernia repair without bowel resection or division of adhesions
* Minor abdominal wound dehiscence unless this causes bowel complications requiring resection
* Non-elective formation of a colostomy or ileostomy as either a trephine or a laparoscopic procedure (NB: if a midline laparotomy is performed, with the primary procedure being formation of a stoma then this should be included)
* Vascular surgery, including abdominal aortic aneurysm repair
* Caesarean section or obstetric laparotomies
* Gynaecological laparotomy
* Ruptured ectopic pregnancy, or pelvic abscesses due to pelvic inflammatory disease
* Laparotomy/laparoscopy for pathology caused by blunt or penetrating trauma
* All surgery relating to organ transplantation (including returns to theatre for any reason following transplant surgery)
* Surgery relating to sclerosing peritonitis
* Surgery for removal of dialysis catheters
* Laparotomy/laparoscopy for oesophageal pathology
* Laparotomy/laparoscopy for pathology of the spleen, renal tract, kidneys, liver, gall bladder and biliary tree, pancreas or urinary tract
* Returns to theatre for complications (eg bowel injury, haematoma, collection) following non-GI surgery are excluded. i.e returns to theatre following renal, urological, gynaecological, vascular, hepatic, pancreatic, splenic surgery are excluded.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Acute general surgical patients presenting with gastrointestinal pathology deemed eligible for NELA who have undergone a diagnostic CT scan of the abdomen (or abdomen and pelvis) who are scheduled to either undergo either operative or non-operative interventions.
Sampling Method: Non-Probability Sample
Enrollment: 294 (Estimated)
Dates: Start 2018-10-01 (Actual); Primary Completion 2019-03-31 (Estimated); Study Completion 2020-08-01 (Estimated)

PRIMARY OUTCOMES:
30-day mortality | 30 days post surgery
  Deaths (all cause) within 30 days of surgical procedure

SECONDARY OUTCOMES:
1 year mortality | 1 year post surgery
  Deaths (all cause) within one year of surgery
Length of stay | Reported at 30 days after surgical procedure
  Index hospital admission length of stay (measured as number of nights as inpatient)
Post-operative morbidity | 30 days post surgery
  Complications following surgery assessed using the Clavien Dindo classification
Destination of discharge from hospital | End of initial hospital inpatient care episode. Closes at time of discharge within 30 days of surgical procedure)
  Place of discharge after hospital care (Home, rehabilitation facility, nursing or care home)
Hospital readmission | 30 days after discharge
  Unplanned readmission to hospital
Participant care needs at time of hospital discharge | End of initial hospital inpatient care episode. Closes at time of discharge within 30 days of surgical procedure)
  Frequency, length and nature of care needs and formal support required to allow safe discharge

CONTACTS AND LOCATIONS:
Overall Officials: Malcolm West, MD PhD MRCS, Principal Investigator — University of Southampton
Locations (10):
- United Kingdom (10):
  - Hampshire Hospitals NHS Foundation Trust, Basingstoke
  - Royal Bournemouth and Christchurch Hospitals NHS Foundation Trust, Bournemouth
  - Dorset County Hospital NHS Foundation Trust, Dorchester
  - Isle of Wight NHS Trust, Newport
  - Poole Hospital NHS Foundation Trust, Poole
  - Portsmouth Hospitals NHS Trust, Portsmouth
  - Salisbury NHS Foundation Trust, Salisbury
  - University Hospital Southampton NHS Foundation Trust, Southampton
  - Hampshire Hospitals NHS Foundation Trust, Winchester
  - Yeovil District Hospital NHS Foundation Trust, Yeovil

IPD SHARING:
Plan to Share IPD: No
No sharing plan